CLINICAL TRIAL: NCT06994195
Title: A Phase III Randomized Controlled Clinical Study Comparing BL-B01D1 With the Investigator's Choice of Chemotherapy in Patients With Platinum-resistant Recurrent Epithelial Ovarian Cancer
Brief Title: A Study Comparing BL-B01D1 With the Investigator's Choice of Chemotherapy in Patients With Platinum-resistant Recurrent Epithelial Ovarian Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-310
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — liposomal doxorubicin; Paclitaxel; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BL-B01D1 (Experimental): Participants receive BL-B01D1 in the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-B01D1
- Investigator's choice of chemotherapy (Active Comparator): Participants receive Liposomal doxorubicin, Paclitaxel or Topotecan in the first cycle (4 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: Liposomal doxorubicin, Paclitaxel or Topotecan

INTERVENTIONS:
Drug: BL-B01D1 — Administration by intravenous infusion for a cycle of 3 weeks.
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507
  Arms: BL-B01D1
Drug: Liposomal doxorubicin, Paclitaxel or Topotecan — Administration by intravenous infusion for a cycle of 4 weeks.
  Arms: Investigator's choice of chemotherapy

SUMMARY:
This trial is a registered, phase III, randomized, open-label, multicenter study to evaluate the efficacy and safety of BL-B01D1 in patients with platinum-resistant recurrent epithelial ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form and comply with the protocol requirements;
2. Age: ≥18 years old;
3. Expected survival time ≥3 months;
4. Histologically or cytologically confirmed epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer;
5. Previously treated with a platinum-based regimen and confirmed to have platinum-resistant recurrence;
6. Previously received 1-3 lines of systemic anti-tumor therapy, with radiographic evidence of disease progression during or after the last line of treatment or intolerance to the current treatment prior to randomization;
7. For subjects with documented folate receptor-alpha (FRα) positivity, progression must have occurred after treatment with mirvetuximab soravtansine;
8. Agree to provide archived tumor tissue specimens or fresh tissue samples from the primary or metastatic lesions within the past 3 years;
9. Must have at least one measurable lesion as defined by RECIST v1.1;
10. ECOG performance status score of 0 or 1;
11. Toxicity from prior anti-tumor therapy has recovered to ≤ Grade 1 as defined by NCI-CTCAE v5.0;
12. No severe cardiac dysfunction, with left ventricular ejection fraction ≥50%;
13. Organ function levels must meet the requirements;
14. Coagulation function: International Normalized Ratio (INR) ≤1.5, and activated partial thromboplastin time (APTT) ≤1.5×ULN;
15. For premenopausal women with childbearing potential, a serum pregnancy test must be performed within 7 days before starting treatment, and the result must be negative; they must not be breastfeeding. All enrolled patients should use adequate barrier contraception throughout the treatment period and for 6 months after treatment ends.

Exclusion Criteria:

1. Use of chemotherapy, targeted therapy, biologic therapy, etc., within 4 weeks or 5 half-lives prior to study randomization and palliative radiotherapy, etc., within 2 weeks;
2. Patients with locally advanced or metastatic platinum-resistant recurrent epithelial ovarian cancer who are eligible for radical locoregional therapy;
3. Front line received ADCs targeting topoisomerase I inhibitors or EGFR and/or HER3;
4. History of severe heart disease and cerebrovascular disease;
5. Unstable thrombotic events requiring therapeutic intervention within 6 months before screening;
6. Prolonged QT interval, complete left bundle branch block, III degree atrioventricular block, frequent and uncontrollable arrhythmia;
7. Diagnosed with active malignancy within 3 years before randomization;
8. Hypertension poorly controlled by two antihypertensive drugs;
9. Patients with poor glycemic control;
10. Patients with grade ≥1 radiation pneumonitis according to the RTOG/EORTC definition; Previous history of ILD;
11. Complicated with pulmonary diseases leading to clinically severe respiratory function impairment;
12. Patients with active central nervous system metastases;
13. Severe infection occurred within 4 weeks before randomization in study 13; Evidence of pulmonary infection or active pulmonary inflammation within 2 weeks before randomization;
14. Patients with massive or symptomatic effusions or poorly controlled effusions;
15. Imaging examination showed that the tumor had invaded or enveloped the large blood vessels in the abdomen, chest, neck, and pharynx;
16. Serious unhealed wound, ulcer or fracture within 4 weeks before signing the informed consent;
17. Subjects with clinically significant bleeding or obvious bleeding tendency within 4 weeks before signing the informed consent;
18. Patients with inflammatory bowel disease, extensive bowel resection, immune enteritis, intestinal obstruction or chronic diarrhea;
19. Patients with a history of allergy to recombinant humanized antibodies or to any of the excipients of BL-B01D1;
20. Had a history of autologous or allogeneic stem cell transplantation;
21. Human immunodeficiency virus antibody positive, active hepatitis B virus infection or hepatitis C virus infection;
22. A history of severe neurological or psychiatric illness;
23. Received other unmarketed investigational drugs or treatments within 4 weeks before randomization;
24. Subjects who were scheduled to be vaccinated or received live vaccine within 28 days before study randomization;
25. Other circumstances in which the investigator considered it inappropriate to participate in the trial because of complications or other circumstances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  Progression-free survival (PFS) as assessed by BIRC is defined as the time between the date subjects are randomized and the first observation of disease progression (based on BICR's image-based assessment) or death.
Overall survival (OS) | Up to approximately 24 months
  Overall survival (OS) is defined as the time between the subject's randomization date and subject's death.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 24 months
  Objective response rate (ORR) is defined as the number of CR and PR in the treatment and control groups divided by the number of that group in the full analysis set (FAS).
Disease Control Rate (DCR) | Up to approximately 24 months
  Disease Control Rate (DCR) : Percentage of all randomized subjects who rated the best overall response (BOR) as complete response (CR), partial response (PR), and disease stabilization (SD) according to RECIST 1.1 criteria.
Duration of Response (DOR) | Up to approximately 24 months
  Duration of Response (DOR) : defined as the period from the date when tumor response is first recorded to the date when objective tumor progression is first recorded or the date of death.
RR (Response Rate) | Up to approximately 24 months
  RR is defined as the proportion of subjects with an overall assessment of remission by RECIST v1.1 and GCIG CA-125 criteria.
CA-125 Response Rate | Up to approximately 24 months
  CA-125 Response Rate is defined as the proportion of subjects evaluated as remission by GCIG CA-125 criteria.
Treatment Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-B01D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-B01D1.
Anti-drug antibody (ADA) | Up to approximately 24 months
  Frequency of anti-BL-B01D1 antibody (ADA) will be investigated.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China